CLINICAL TRIAL: NCT04501380
Title: A Randomized Open Label Trial Evaluating the Efficacy of AEMCOLO (Rifamycin SV MMX) in the Treatment of Small Intestinal Bacterial Overgrowth (SIBO)
Brief Title: Efficacy of AEMCOLO (Rifamycin SV MMX) in the Treatment of Small Intestinal Bacterial Overgrowth (SIBO)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bradley Connor (Other)
Responsible Party: Sponsor-Investigator, Bradley Connor, Principal Investigator, The New York Center for Travel and Tropical Medicine
Organization: The New York Center for Travel and Tropical Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAS 0519-1
Record Dates: First submitted 2020-07-28; First posted 2020-08-06 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Small Intestinal Bacterial Overgrowth; Gastrointestinal Disease; Gastrointestinal Infection
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — rifamycin SV

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1st regimen (Experimental): 15 patients will receive AEMCOLO (Rifamycin SV MMX) 194 mg two tablets to take twice daily for 14 days (56 Tablets)
  Interventions: Drug: AEMCOLO (Rifamycin SV MMX)
- 2nd regimen (Experimental): 15 patients will receive AEMCOLO (Rifamycin SV MMX) 194 mg tablets to take two tablets three times daily for 14 days (84 Tablets).
  Interventions: Drug: AEMCOLO (Rifamycin SV MMX)

INTERVENTIONS:
Drug: AEMCOLO (Rifamycin SV MMX) — Participants will be issued a patient kit containing AEMCOLO (Rifamycin SV MMX) 194 mg tablets for the 1st or the 2nd treatment regimen in a random order.

SUMMARY:
Open label interventional randomized pilot study utilizing two dosing regimens of AEMCOLO. The goal of this study is to evaluate effectiveness of a novel antibiotic, AEMCOLO (Rifamycin SV MMX) in the treatment of Small intestinal bacterial overgrowth (SIBO).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms compatible with SIBO
* A positive breath test for either hydrogen predominant, methane predominant or mixed SIBO

Exclusion Criteria:

* History of diabetes mellitus,
* Diarrhea predominant irritable bowel syndrome (IBS-D),
* Symptomatic bowel obstruction,
* Diverticulitis and/ or adhesions,
* Autoimmune disorder,
* Immunosuppression by medication or disease,
* Pregnant or breast feeding,
* The use of antibiotics, probiotics or prebiotics within the previous 30 days,
* Known hypersensitivity to rifamycin, any of the other rifamycin class antimicrobial agents (e.g. rifaximin), or any of the components of AEMCOLO.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the change of an abnormal breath test followed by a regimen of AEMCOLO | 1 month after treatment
  A hydrogen and methane breath test will be used to measure presence or absence of Small Intestinal Bacterial Overgrowth (SIBO). Study subjects will be assessed for the presence of SIBO. A rise of ≥ 20 ppm from baseline in hydrogen by 90 minutes or a level of ≥ 10 ppm for methane is considered a positive test for SIBO on a breath test. When combining both hydrogen and methane in the breath test, a rise of ≥ 15 ppm from baseline at 90 minutes is considered a positive test for SIBO. We plan to measure these parameters at baseline and after completion of study medication.

SECONDARY OUTCOMES:
To evaluate the change in clinical symptoms followed by a regimen of AEMCOLO | Daily survey during and after treatment for 2 months and follow up at 3 months
  There will be a measurement of symptoms as assessed by a validated visual analogue scale (VAS) questionnaire. Symptoms will be assessed on a 0-4 scale to generate a maximum score of 20 and a minimum score of 0. The change in this composite score will be compared between two treatment arms at baseline, after completion of study medication, and 3 months after treatment. A positive clinical response defined as a 50% reduction in CS will be assessed. This method of analysis closely follows the multinational consensus recommended guidelines for data analysis in IBS clinical studies.

CONTACTS AND LOCATIONS:
Locations (1):
- The New York Center for Travel and Tropical Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dukowicz AC, Lacy BE, Levine GM. Small intestinal bacterial overgrowth: a comprehensive review. Gastroenterol Hepatol (N Y). 2007 Feb;3(2):112-22. PMID 21960820
- [Background] Quigley EM, Abu-Shanab A. Small intestinal bacterial overgrowth. Infect Dis Clin North Am. 2010 Dec;24(4):943-59, viii-ix. doi: 10.1016/j.idc.2010.07.007. PMID 20937459
- [Background] Sachdev AH, Pimentel M. Gastrointestinal bacterial overgrowth: pathogenesis and clinical significance. Ther Adv Chronic Dis. 2013 Sep;4(5):223-31. doi: 10.1177/2040622313496126. PMID 23997926
- [Background] Shah SC, Day LW, Somsouk M, Sewell JL. Meta-analysis: antibiotic therapy for small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2013 Oct;38(8):925-34. doi: 10.1111/apt.12479. Epub 2013 Sep 4. PMID 24004101
- [Background] Pimentel M, Chang C, Chua KS, Mirocha J, DiBaise J, Rao S, Amichai M. Antibiotic treatment of constipation-predominant irritable bowel syndrome. Dig Dis Sci. 2014 Jun;59(6):1278-85. doi: 10.1007/s10620-014-3157-8. Epub 2014 May 1. PMID 24788320
- [Background] Gatta L, Scarpignato C. Systematic review with meta-analysis: rifaximin is effective and safe for the treatment of small intestine bacterial overgrowth. Aliment Pharmacol Ther. 2017 Mar;45(5):604-616. doi: 10.1111/apt.13928. Epub 2017 Jan 12. PMID 28078798
- [Background] Rezaie A, Buresi M, Lembo A, Lin H, McCallum R, Rao S, Schmulson M, Valdovinos M, Zakko S, Pimentel M. Hydrogen and Methane-Based Breath Testing in Gastrointestinal Disorders: The North American Consensus. Am J Gastroenterol. 2017 May;112(5):775-784. doi: 10.1038/ajg.2017.46. Epub 2017 Mar 21. PMID 28323273
- [Background] Pimentel M, Chow EJ, Lin HC. Normalization of lactulose breath testing correlates with symptom improvement in irritable bowel syndrome. a double-blind, randomized, placebo-controlled study. Am J Gastroenterol. 2003 Feb;98(2):412-9. doi: 10.1111/j.1572-0241.2003.07234.x. PMID 12591062
- [Background] Furnari M, Parodi A, Gemignani L, Giannini EG, Marenco S, Savarino E, Assandri L, Fazio V, Bonfanti D, Inferrera S, Savarino V. Clinical trial: the combination of rifaximin with partially hydrolysed guar gum is more effective than rifaximin alone in eradicating small intestinal bacterial overgrowth. Aliment Pharmacol Ther. 2010 Oct;32(8):1000-6. doi: 10.1111/j.1365-2036.2010.04436.x. Epub 2010 Aug 18. PMID 20937045
- [Background] Ghoshal UC, Ghoshal U, Das K, Misra A. Utility of hydrogen breath tests in diagnosis of small intestinal bacterial overgrowth in malabsorption syndrome and its relationship with oro-cecal transit time. Indian J Gastroenterol. 2006 Jan-Feb;25(1):6-10. PMID 16567886
- [Derived] Connor BA, Rogova M, Garcia J, Gardner M, Waraich C, Averill V. A randomized open label pilot study evaluating the efficacy of two dosing regimens of rifamycin SV MMX in the treatment of small intestinal bacterial overgrowth. BMC Gastroenterol. 2025 Apr 3;25(1):219. doi: 10.1186/s12876-025-03804-3. PMID 40181268